CLINICAL TRIAL: NCT04145921
Title: Effectiveness of Fast-track Clinical Pathway on Minimally-invasive Total Hip Arthroplasty Surgery in NTUH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201207008RIC
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS for MIS-THA (Experimental): enhanced recovery after surgery (ERAS) pathway for minimally-invasive surgery of total hip arthroplasty (MIS-THA)
  Interventions: Procedure: ERAS for MIS-THA
- conventional MIS-THA (Active Comparator): conventional pathway for minimally-invasive surgery of total hip arthroplasty (MIS-THA)
  Interventions: Procedure: conventional MIS-THA

INTERVENTIONS:
Procedure: ERAS for MIS-THA — enhanced recovery after surgery (ERAS) pathway for minimally-invasive surgery of total hip arthroplasty (MIS-THA)
  Arms: ERAS for MIS-THA
Procedure: conventional MIS-THA — conventional pathway for minimally-invasive surgery of total hip arthroplasty (MIS-THA)
  Arms: conventional MIS-THA

SUMMARY:
The objective of this study was to evaluate the effects of an enhanced recovery after surgery (ERAS) pathway incorporated with pre-operative physical therapy and education on immediate and short-term outcomes of minimally-invasive surgery of total hip arthroplasty (MIS-THA). We hypothesized that this ERAS pathway can shorten post-operative length of hospital stay and ensure same-day independent mobilization in MIS-THA. The first specific aim was to compare primary immediate outcomes, including post-operative length of hospital stay and the rate of same-day independent mobilization, between ERAS for MIS-THA patients and conventional MIS-THA patients. The second aim was to compare other immediate outcomes, including post-operative pain scores, analgesics usage, the rate of blood transfusion and post-operative nausea and vomiting (PONV), between the two groups of patients. Third, we aimed to compare short-term outcomes, including post-operative 1-year Harris hip score, Oxford hip score and EQ-5D index of quality of life, between the two groups of patients. We also compared hospital cost and profit between the two groups of patients. Moreover, we identified the factors affecting post-operative length of hospital stay in ERAS for MIS-THA patients.

DETAILED DESCRIPTION:
Study subjects:

We conducted a prospective comparative study to investigate 50 patients receiving an ERAS pathway incorporated with pre-operative physical therapy and education for MIS-THA and 25 patients receiving conventional MIS-THA. We included the patients with advanced osteonecrosis of femoral head or hip osteoarthritis receiving unilateral primary MIS-THA performed by the same surgeon at the same hospital. We excluded patients with renal or hepatic function impairment which precluded multimodal pain control. However, we did not preselect patients with younger age or better activity level. This study was approved by the Institutional Review Board at National Taiwan University Hospital. Written informed consent was obtained from all patients.

ERAS for MIS-THA versus conventional MIS-THA:

In this study, ERAS for MIS-THA was defined as the ERAS pathway incorporated with pre-operative short-term physical therapy and education for MIS-THA. On the other hand, conventional MIS-THA in this study was defined as the conventional pathway without pre-operative physical therapy and education for MIS-THA. Both of ERAS for MIS-THA and conventional MIS-THA comprised the same MIS-THA techniques, multimodal pain control, standardized volume management and PONV prophylaxis, deep vein thrombosis prophylaxis and post-operative rehabilitation program.

Pre-operative physical therapy and education:

Pre-operatively in the outpatient clinics, we informed patients that the discharge days depended on the rehabilitation progress by oral and written information. We also gave patients the detailed information about rehabilitation program and discharge criteria. We consulted physical therapy specialists for one session of physical therapy intervention before operation. The standardized pre-operative physical therapy programs included three parts. First, posterior dislocation precautions were well explained to the patients, including no hip flexion greater than 90 degrees, no hip adduction or hip internal rotation beyond neutral, and no combination of the above motions. Then, therapeutic exercise programs given in acute post-operative inpatient phase were demonstrated and practiced, including ankle pumps, quadriceps sets, gluteal sets, bed-supported knee bends, active hip abduction, and straight leg raising. The patients were instructed to do these exercises by themselves at home until the day of operation. Last, the patients received activity and functional training, including bed mobility, transfer skills, gait training with appropriate assistive device and weight bearing to tolerance, stair training, and modified activities of daily living following precautions.

MIS-THA techniques:

We utilized posterolateral mini-incision techniques with posterior capsulotendinous repair to the posterolateral aspect of greater trochanter bone for every patient receiving MIS-THA. The incision size was routinely 5-8 cm with hip in flexion position based on body build. We did not use surgical drains.

Multimodal pain control:

For post-operative analgesia, we used multimodal pain control protocols including pre-emptive oral analgesics (acetaminophen, celecoxib, tramadol, gabapentin), intra-operative periarticular injection with cocktail mix of analgesics and antibiotics (levobupivacaine, ketorolac, epinephrine, cefazolin), post-operative oral analgesics (acetaminophen, celecoxib, tramadol, gabapentin), and intramuscular ketorolac as needed to control pain without reliance on morphine. Levobupivacaine used in our periarticular injection is a safer analgesic compared with bupivacaine in terms of cardiovascular adverse effects. We did not routinely use patient-controlled analgesia (PCA) pumps containing morphine unless there was a request from the patient.

Standardized volume management and PONV prophylaxis:

For standardized volume management, we used tetrastarch colloid solutions and restrictive strategy of allogenic blood transfusion (hemoglobin < 9 g/dl with altered vital signs or hemoglobin < 7 g/dl without altered vital signs). For PONV prophylaxis and treatment, we used esomeprazole, metoclopramide, ondansetron, and normovolemic fluid control with tetrastarch colloid solutions.

Deep vein thrombosis prophylaxis:

For deep vein thrombosis prophylaxis, we used anti-embolism stockings and daily enoxaparin (40mg) starting from 12 hours after operation for 2 days then oral aspirin for 6 weeks. We used a short-duration anti-thrombotic agent combined with aspirin and early mobilization because the risk of deep vein thrombosis after THA with short-duration pharmacological prophylaxis and early mobilization was quite low. Besides, Asians have a 70% lower prevalence of venous thromboembolism compared to Caucasians.

Post-operative rehabilitation program:

Post-operative rehabilitation program was the same as pre-operative physical therapy and was conducted with close observation of patient's pain tolerance and general conditioning. All patients were discharged direct to their residences without any home-care rehabilitation service.

Discharge criteria:

For ERAS for MIS-THA patients and conventional MIS-THA patients, we used uniform discharge criteria including being self-dependent, being able to walk with crutches or walkers, sufficient pain control with oral analgesics, no infection signs, well knowledge of position restriction, and being able to perform home exercise.

Outcome measures:

A database was established for prospective collection of patient demographic, pre- and post-operative data for statistical analysis. The evaluator was blinded to the grouping of patients in data collection. Primary immediate outcomes were post-operative length of hospital stay and the rate of same-day independent mobilization (ambulation without assistance from another person within 24 hours after operation). Other immediate outcomes included post-operative visual analog scale (VAS) pain scores, analgesics usage, the rate of blood transfusion and PONV. Short-term outcomes were post-operative 1-year Harris hip score, Oxford hip score, and EQ-5D index of self-reported health-related quality of life. We also recorded adverse events as well as hospital cost and profit.

Statistical analysis:

A priori sample size determination was based on post-operative length of hospital stay, which was the primary outcome measure. The sample size was calculated to detect a mean difference of 3 days in post-operative length of stay between ERAS for MIS-THA patients and conventional MIS-THA patients assuming a standard deviation of 3.5 days. We assumed a two-sided type I error of 0.05 and a power of 80%. This resulted in a required sample size of 22 in each group. In this study, we included 50 patients in ERAS group and 25 patients in conventional group, respectively. The case number in this study was sufficient for a priori sample size calculation.

Data are presented as mean ± standard deviation and ratio. Student t-test, Mann-Whitney U test, Chi-square test and Fisher exact test were used to compare continuous or categorical variables between different groups of subjects. Multivariable regression analysis by best subset regression was used to identify significant variables affecting post-operative length of hospital stay. Longitudinal analysis by Generalized Estimating Equations (GEE) using robust standard errors was used to compare repeated measurements such as post-operative VAS pain scores. STATA 11 statistical software (StataCorp LP, College Station, TX, USA) was used for statistical analysis. A two-tailed p value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with advanced osteonecrosis of femoral head or hip osteoarthritis receiving unilateral primary minimally-invasive surgery of total hip arthroplasty (MIS-THA) performed by the same surgeon at the same hospital

Exclusion Criteria:

* patients with renal or hepatic function impairment which precluded multimodal pain control

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
post-operative length of hospital stay | up to 2 weeks after operation
  post-operative length of hospital stay
rate of same-day independent mobilization | up to 24 hours after operation
  rate of same-day independent mobilization (ambulation without assistance from another person within 24 hours after operation)

SECONDARY OUTCOMES:
post-operative VAS pain scores | up to 24 hours after operation
  post-operative visual analog scale (VAS) pain scores
post-operative analgesics usage | up to 2 weeks after operation
  post-operative analgesics usage
the rate of blood transfusion | up to 2 weeks after operation
  the rate of blood transfusion
rate of PONV | up to 2 weeks after operation
  rate of post-operative nausea and vomiting (PONV)
post-operative 1-year Harris hip score | 1 year after operation
  post-operative 1-year Harris hip score
post-operative 1-year Oxford hip score | 1 year after operation
  post-operative 1-year Oxford hip score
post-operative 1-year EQ-5D index of quality of life | 1 year after operation
  post-operative 1-year EQ-5D index of self-reported health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Ti Wang, MD,PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No